CLINICAL TRIAL: NCT01745107
Title: Phase Ⅲ Study of Prophylactic Postoperative Intensity Modulated Radiation Therapy in Stage T2-3N0M0 Disease of Thoracic Esophageal Squamous Cell Carcinoma;
Brief Title: Efficacy of Intensity Modulated Radiation Therapy After Surgery in Early Stage of Esophageal Carcinoma;
Acronym: IMRT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Sichuan Cancer Hospital and Research Institute (Other); Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Zefen Xiao, Clinical Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z121107001012004; Z121107001012004 (Other: Beijing Municipal Science & Technology Commission,China)
Record Dates: First submitted 2012-12-06; First posted 2012-12-07 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Esophageal Neoplasm; Esophageal Cancer TNM Staging Primary Tumor (T) T2; Esophageal Cancer TNM Staging Primary Tumor (T) T3; Esophageal Cancer TNM Staging Regional Lymph Nodes (N) N0; Esophageal Cancer TNM Staging Distal Metastasis (M) M0
Keywords: T2-3N0M0 disease of esophageal neoplasm; postoperative radiotherapy; intensity modulated radiation therapy; survival
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgery alone (No Intervention): No prophylactic postoperative radiation therapy,that is surgery alone is developed in this arm
- surgery plus radiation (Experimental): Prophylactic postoperative radiation therapy is developed in this arm
  Interventions: Radiation: Prophylactic postoperative radiation therapy

INTERVENTIONS:
Radiation: Prophylactic postoperative radiation therapy — Prescription dose of 95%planning target volume(PTV) 50.4Gy/1.8Gy/28fractions for supraclavicular region and 95%PTV 56Gy/2Gy/28fractions for mediastinum which is delivered in 2 months after surgery.
  Other Names: Preventive postoperative radiotherapy
  Arms: surgery plus radiation

SUMMARY:
The purpose of this study is to determine the efficacy of preventive intensity modulated radiation therapy after surgery in stage T2-3N0M0 disease of thoracic esophageal squamous cell carcinoma(UICC 7th edition) and to identify the subgroup benefiting from the treatment.

DETAILED DESCRIPTION:
Although preoperative chemoradiation therapy followed by surgery is the most common approach for patients with resectable esophageal cancer, the considerable number of esophageal cancer patients received operation as the first treatment modality. Accordingly, postoperative treatments have been playing an important role because of the poor survival rates of the patients who have been treated with resection alone. The existing data shows that the 5-yeal survival rate of stage T2-3N0M0(UICC 7th edition) of thoracic esophageal squamous cell carcinoma(TESCC) after surgery is about 50% ,and locoregional lymph nodes metastases is responsible for the main cause of failure while distal metastases account for relatively less ratio. Therefore, the subclinical residual tumor is affirmative even if the early disease has been undergone curable excision and local adjuvant treatment may be essential. While we have proved the value of prophylactic radiation therapy after radical esophagectomy for esophageal carcinoma with positive lymph node metastases and stage Ⅲ disease, there is still lack of clear evidence for prophylactic radiation therapy in stage T2-3N0M0 disease now. The comparison of conventional 2-dimensional radiotherapy after operation versus surgery alone does not show statistically significant difference for stage T2-3N0M0 disease in our previous report. In the precise radiotherapy setting, more and more evidences of non-randomised control study indicate the trend or preliminary results of dosimetric advantages of IMRT translating into substantive benefits in both survival and locoregional control compared with 3- dimensional conformal and 2-dimensional conventional radiotherapy for the treatment of esophageal carcinoma, but it remains to be confirmed in the randomized control study that whether the IMRT is effective to improve the clinical outcomes of stage T2-3N0M0 patients of TESCC. In view of this, we designed the randomized controlled trial to determine the clinical efficacy and toxicity of prophylactic IMRT after surgery in stage T2-3N0M0 disease of TESCC.

ELIGIBILITY:
Inclusion Criteria:

* Stage T2-3N0M0 disease of TESCC patients confirmed by pathology studies who received R0 operations in Cancer Institute & Hospital，CAMS；
* KPS≥70 before radiotherapy;
* Did not receive neoadjuvant or adjuvant treatment;
* No clear recurrent or metastatic lesions before radiotherapy;
* Intensity modulated radiation therapy(IMRT) is accepted;
* Regular follow-up.

Exclusion Criteria:

* Exploratory thoracotomy or palliative surgery;
* No clear recurrent or metastatic sites;
* Recurrence or metastasis is not certain;
* death of no definite cause.
* Irregular follow-up;

Ages: 40 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival time | up to 3 years
  including survival time from randomization to locoregional recurrence and to distal metastasis

SECONDARY OUTCOMES:
overall survival time | up to 5 years
  survival time from randomization to death

CONTACTS AND LOCATIONS:
Overall Officials: Zefen Xiao, MD, Principal Investigator — The Department of Radiation Oncology ,Cancer Institute & Hospital，Chinese Academy of Medical Science
Locations (1):
- Cancer institute & Hospital，Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Xiao ZF, Yang ZY, Liang J, Miao YJ, Wang M, Yin WB, Gu XZ, Zhang DC, Zhang RG, Wang LJ. Value of radiotherapy after radical surgery for esophageal carcinoma: a report of 495 patients. Ann Thorac Surg. 2003 Feb;75(2):331-6. doi: 10.1016/s0003-4975(02)04401-6. PMID 12607634
- [Background] Lin SH, Wang L, Myles B, Thall PF, Hofstetter WL, Swisher SG, Ajani JA, Cox JD, Komaki R, Liao Z. Propensity score-based comparison of long-term outcomes with 3-dimensional conformal radiotherapy vs intensity-modulated radiotherapy for esophageal cancer. Int J Radiat Oncol Biol Phys. 2012 Dec 1;84(5):1078-85. doi: 10.1016/j.ijrobp.2012.02.015. Epub 2012 Aug 3. PMID 22867894
- [Background] Chen J, Zhu J, Pan J, Zhu K, Zheng X, Chen M, Wang J, Liao Z. Postoperative radiotherapy improved survival of poor prognostic squamous cell carcinoma esophagus. Ann Thorac Surg. 2010 Aug;90(2):435-42. doi: 10.1016/j.athoracsur.2010.04.002. PMID 20667325
- [Background] Mariette C, Balon JM, Piessen G, Fabre S, Van Seuningen I, Triboulet JP. Pattern of recurrence following complete resection of esophageal carcinoma and factors predictive of recurrent disease. Cancer. 2003 Apr 1;97(7):1616-23. doi: 10.1002/cncr.11228. PMID 12655517
- [Background] Nishimaki T, Suzuki T, Suzuki S, Kuwabara S, Hatakeyama K. Outcomes of extended radical esophagectomy for thoracic esophageal cancer. J Am Coll Surg. 1998 Mar;186(3):306-12. doi: 10.1016/s1072-7515(98)00013-1. PMID 9510261
- [Background] Reeh M, Nentwich MF, von Loga K, Schade J, Uzunoglu FG, Koenig AM, Bockhorn M, Rosch T, Izbicki JR, Bogoevski D. An attempt at validation of the Seventh edition of the classification by the International Union Against Cancer for esophageal carcinoma. Ann Thorac Surg. 2012 Mar;93(3):890-6. doi: 10.1016/j.athoracsur.2011.11.035. Epub 2012 Jan 29. PMID 22289905
- [Background] Isono K, Sato H, Nakayama K. Results of a nationwide study on the three-field lymph node dissection of esophageal cancer. Oncology. 1991;48(5):411-20. doi: 10.1159/000226971. PMID 1745490
- [Background] Akiyama H, Tsurumaru M, Udagawa H, Kajiyama Y. Radical lymph node dissection for cancer of the thoracic esophagus. Ann Surg. 1994 Sep;220(3):364-72; discussion 372-3. doi: 10.1097/00000658-199409000-00012. PMID 8092902
- [Background] Chen J, Sang M, Chen Y. [Recurrence pattern and prognosis of esophageal cancer following tumor resection]. Zhonghua Zhong Liu Za Zhi. 1998 Jul;20(4):293-5. Chinese. PMID 10920988
- [Background] Visbal AL, Allen MS, Miller DL, Deschamps C, Trastek VF, Pairolero PC. Ivor Lewis esophagogastrectomy for esophageal cancer. Ann Thorac Surg. 2001 Jun;71(6):1803-8. doi: 10.1016/s0003-4975(01)02601-7. PMID 11426751
- [Background] Teniere P, Hay JM, Fingerhut A, Fagniez PL. Postoperative radiation therapy does not increase survival after curative resection for squamous cell carcinoma of the middle and lower esophagus as shown by a multicenter controlled trial. French University Association for Surgical Research. Surg Gynecol Obstet. 1991 Aug;173(2):123-30. PMID 1925862
- [Background] Fok M, Sham JS, Choy D, Cheng SW, Wong J. Postoperative radiotherapy for carcinoma of the esophagus: a prospective, randomized controlled study. Surgery. 1993 Feb;113(2):138-47. PMID 8430362
- [Background] Zieren HU, Muller JM, Jacobi CA, Pichlmaier H, Muller RP, Staar S. Adjuvant postoperative radiation therapy after curative resection of squamous cell carcinoma of the thoracic esophagus: a prospective randomized study. World J Surg. 1995 May-Jun;19(3):444-9. doi: 10.1007/BF00299187. PMID 7639004
- [Background] Chen G, Wang Z, Liu XY, Liu FY. Recurrence pattern of squamous cell carcinoma in the middle thoracic esophagus after modified Ivor-Lewis esophagectomy. World J Surg. 2007 May;31(5):1107-14. doi: 10.1007/s00268-006-0551-1. PMID 17426905
- [Background] Xiao ZF, Yang ZY, Miao YJ, Wang LH, Yin WB, Gu XZ, Zhang DC, Sun KL, Chen GY, He J. Influence of number of metastatic lymph nodes on survival of curative resected thoracic esophageal cancer patients and value of radiotherapy: report of 549 cases. Int J Radiat Oncol Biol Phys. 2005 May 1;62(1):82-90. doi: 10.1016/j.ijrobp.2004.08.046. PMID 15850906
- [Background] Chen J, Pan J, Zheng X, Zhu K, Li J, Chen M, Wang J, Liao Z. Number and location of positive nodes, postoperative radiotherapy, and survival after esophagectomy with three-field lymph node dissection for thoracic esophageal squamous cell carcinoma. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):475-82. doi: 10.1016/j.ijrobp.2010.08.037. Epub 2010 Oct 8. PMID 20934269
- [Background] Bedard EL, Inculet RI, Malthaner RA, Brecevic E, Vincent M, Dar R. The role of surgery and postoperative chemoradiation therapy in patients with lymph node positive esophageal carcinoma. Cancer. 2001 Jun 15;91(12):2423-30. PMID 11413534
- [Background] Qiao XY, Wang W, Zhou ZG, Gao XS, Chang JY. Comparison of efficacy of regional and extensive clinical target volumes in postoperative radiotherapy for esophageal squamous cell carcinoma. Int J Radiat Oncol Biol Phys. 2008 Feb 1;70(2):396-402. doi: 10.1016/j.ijrobp.2007.06.031. Epub 2007 Sep 12. PMID 17855004
- [Background] Zhang Wencheng,Wang Qifeng,Xiao Zefen,et al.A efficacy analysis of intensity-modulated radiotherapy or three-dimensional conformal radiotherapy for resected thoracic esophageal squamous cell carcinoma.Chinese Journal of Radiation Oncology.2012,21(2):136-139.DOI:10.3760/cma.j.issn.1004-4221.2012.02.012.
- See also: It is a national center for cancer research and treatment. It is one of the clinical trial bases approved by the Food and Drug Administration of State (SFDA) — http://www.cicams.ac.cn